CLINICAL TRIAL: NCT04685577
Title: A Randomized, Placebo Controlled, Double-Blind, Single Dose Study To Evaluate The Safety And Tolerability Of Cream In Burn Patients With Induced Dermal Incisions
Brief Title: Safety, Tolerability and Efficacy of Nefopam Cream in Burn Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NEFOPAM-1; W81XWH-19-2-0048 (Other Grant/Funding Number: Department of Defense (DOD)); CDMRP-MB170036 (Other Grant/Funding Number: DOD/Congressionally Directed Medical Research Programs)
Record Dates: First submitted 2020-11-16; First posted 2020-12-28 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Burn; Multiple Body Regions, Max. Second Degree; Third-Degree Burn; Burn Degree Second
Keywords: Hypertrophic scar, Nefopam,Burn patients.
MeSH Terms: conditions — Burns; Cicatrix, Hypertrophic | interventions — Nefopam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: As this is a 2 arm study. One is experimental drug and other is placebo control. No one will know which side of body part having drug and/or placebo. If required, it will be find out but this study is designed as a double blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nefopam (Experimental): NEFOPAM 3% cream will be applied topically to healing deep dermal scratches in the lateral hip of burn patients daily (twice) for 3 weeks during the proliferative phase of wound healing.
  Interventions: Drug: Nefopam
- Placebo (Placebo Comparator): This will work as a placebo for the experimental drug.
  Interventions: Other: Placebo (Vehicle)

INTERVENTIONS:
Drug: Nefopam — Nefopam HCl inhibits the proliferation and viability of human mesenchymal fibroblasts with elevated β-catenin expression without affecting normal fibroblasts. Nefopam HCl primarily targets cells in which β-catenin is above normal physiologic levels. This threshold effect makes Nefopam HCl a good prospective therapeutic agent by limiting its effect to abnormal mesenchymal cells.Nefopam HCl has been found safe and effective for the reduction of dermal scarring following standardized human dermal wounds of critical depth that produces HTS in normal human volunteers Phase 1 study. In the current study, it is proposed that the concentration of the cream will be 3% and the timing of application will be delayed until after re-epithelialization at about 21 days to maximize the antiproliferative effects of NEFOPAM during the fibrotic/proliferative phase of healing.
  Other Names: Nefopam-HCl
  Arms: Nefopam
Other: Placebo (Vehicle) — Participants will receive vehicle with out the investigational product
  Arms: Placebo

SUMMARY:
Burn patients very commonly develop abnormal scars after injury which can be red, raised or elevated, painful and very itchy. They can prevent normal movement of hands and other joints and lead to ugly deformities which makes physical and psychological recovery very difficult. This proposal seeks to test the usefulness of a cream called Nefopam to prevent and treat these bad scars after burns and other injury to the skin. Nefopam is a drug that has been used as a pain medicine in Europe but has been found to have anti-scarring properties in rats and pigs. It has been tested in healthy people and found to be well tolerated and safe. The study purposes to make a scratch in the hip skin in 60 adult burn patients at two burn unit sites, the University of Alberta and the University of California at Davis, Sacramento CA. Burn patients in the study will have a scratch wound in the skin of the each side of the hip, part way through the thickness of the skin which is shallow at first but gets deeper. This scratch is made with a special guide which precisely controls the length and depth of the scratch so that each scratch is the same. Part of the scratch heals without scar and the deeper part heals with a red raised scar over a small region less than 2 inches long. One side will be treated with the drug and the other with a control or placebo are in a white cream that is indistinguishable, where you cannot tell which side contains the drug. Once the wound is nearly healed, usually less than 21 days, the cream will be applied twice daily for three weeks. Measurements will be done about once per month for four months where the healing scratches will be photographed, measurements of the thickness made with ultrasound and mexameter for scar color or pigment and redness. Ultrasound is a painless probe that uses sound waves to measure scar thickness and mexameter is a painless probe on the surface of the scratch to measure color and redness. Both measurements take only minutes to complete. Patients will be asked to answer a scar assessment form about on how they feel each scratch during the treatment and the research staff will also the complete scar form as well. It is the aim of the study to find a cream the works to prevent and reduce scarring after burn injury in military or civilian patients. In the future, an useful cream for scarring in burn patients may also be helpful for other skin damage which leads to scarring.

DETAILED DESCRIPTION:
Background:

Fibroproliferative disorders (FPD) are common and serious disorders involving many human tissues and are a leading cause of mortality and reported as high a 45% of annual deaths. Hypertrophic scar (HTS) and keloids are the dermal equivalent of FPD and impose lower mortality but great morbidity, particularly following burn injury. In the US, 1.25 million people are treated for burns annually, 50,000 requiring hospitalization. Although the mortality rate for burn injury has improved, burn patients experience a prolonged hospitalization (mean 26.2 days) and rehabilitation, requiring an average of 12.7 weeks off work for patients with thermal injuries >30% of the TBSA. Much of the rehabilitation relates to functional and cosmetic limitations imposed by HTS, including a reduction in range of motion of the extremities and the intense pruritus and heat intolerance making early return to work prohibitive, until remodelling of the HTS has occurred. Although risk factors for HTS include sex, age, racial or genetic factors, and wound location, HTS develops after prolonged inflammation of slowly healing burn wounds with a very high frequency especially in deep dermal wounds independent of other factors in up to 75% of burn patients. Unfortunately, HTS and keloid are known to respond poorly to current forms of therapy, including pressure garments, topically applied silicone and intralesional steroids, usually slowly over months or years, often incompletely. Advances in the immunology of FPD including HTS and keloids, reveal many common features, such that novel advances in therapy for these disorders may provide far reaching benefits to many patients and military personnel suffering from severe scarring after burn injury.

Drug Information: NEFOPAM HCL has been found safe and effective for the reduction of dermal scarring following standardized human dermal wounds of critical depth that produces HTS in normal human volunteers. NEFOPAM HCl was first developed as a non-narcotic analgesic drug and it is currently marketed primarily in Europe, New Zealand and parts of Asia for oral, intramuscular or intravenous use for acute or chronic pain. NEFOPAM HCl has over 30 years of human safety data. It is considered generally safe with mild side effects including nausea, sweating, dry mouth and tachycardia. NEFOPAM reformulated into a cream and topically administered has been shown to reduce the amount of scar tissue formed during wound healing in mice and the red Duroc pig model of hypertrophic scarring. Most recently, a phase I safety and efficacy study was conducted in human volunteers using a standardized progressively deeper dermal wound (0-1.6 mm in depth over 6 cm) made with a sterile jig in each hip, where normotrophic (negative control) and HTS (positive control) develop in the superficial and deep regions of the scratch. 24 patients have been studied over 104 days where the preliminary results demonstrate that NEFOPAM cream has very few adverse side effects, low immunogenicity and encouraging antifibrotic effects on the healing wounds.

Purpose/ Hypothesis:

To re-assess the safety, local tolerability and efficacy of NEFOPAM Cream in burn patients when applied to bilateral deep dermal wounds using a standardized dermal scratch model of hypertrophic scarring.

Objectives:

To assess the efficacy of NEFOPAM Cream versus placebo (vehicle) in reducing scar size following artificially induced dermal wounds in each lateral hip region of burn patients.

To determine the efficacy on wound closure of NEFOPAM Cream versus placebo (vehicle) in burn patients.

To assess the satisfaction of burn patients and investigators in the scar rating and appearance after topical application of NEFOPAM Cream versus placebo (vehicle).

To determine the efficacy of NEFOPAM Cream versus placebo on the gene and protein expression of fibrotic molecules including type I and type III collagen, β-catenin target gene (AXIN-2), TGF- β1, and decorin, quantitative measures of collagen orientation index (COI), immunohistochemistry of a-SMA (smooth muscle actin) and β -catenin in scar tissue.

Research Method/Procedures:

This study will be a double blind, placebo-controlled, randomized multicenter Phase II study in which burn patients will be randomized to receive NEFOPAM Cream or placebo. Qualifying subjects will be randomized to receive 2.0 mL of NEFOPAM Cream or placebo (vehicle) on Day -1 on intact skin in an area on the upper hip not intended for the incision. On Day 0 burn patients who are free of adverse events will enter the treatment phase of the study.

Consenting burn patients requiring skin graft surgery will be scratch-wounded under aseptic conditions on the lateral hip of each lower extremity while under local anesthesia or general anesthesia for their wound debridement as previously described. To create small standardized depth uniform wounds, a jig fitted with a sterile No.11 surgical scalpel blade will be used to create a wound that is 6 cm in length and from 0 to approximately 1.6 mm maximum depth into the deep dermis of the lateral hip mid-distance between the anterior superior iliac spine and the lateral trochanter of the hip. Two identical wounds will be made, one on each hip and subjects will be randomized to receive treatment with NEFOPAM Cream or placebo on each wound. Wounds will be followed until >90% re-epithelialized before the wounds will be cleaned and the cream will be applied twice a day for the next 21 days. The wounds will be covered with an occlusive dressing until Day 21 of treatment (Tegaderm ™). Once the treatment is completed and the wounds are fully healed, the wound/scar will be left uncovered and treated with a moisturizing cream (Glaxal™) if necessary.

Burn patients randomized to receive active treatment will have one wound treated with NEFOPAM Cream (treatment wound site) and the other wound site treated with placebo cream/vehicle (control wound site) according to the randomization schedule and dosing instructions. All study team members and subjects will be blinded to all treatments.

Subjects will receive two applications of treatment to each wound per day for 21 days after the wounds are 90% healed.

Wound evaluations will be performed daily through the treatment period. Digital photography of the wound/scar will occur following wounding and on Day 6 (+/- 2), Day 13 (+/- 2), Day 20 (+/- 3), Day 27 (+/- 2), Day 48 (+/- 7) Day 76 (+/-14), Day 104 (+/- 15). Modified VBSA and POSAS scale, vascularity and pigmentation via Mexameter® and ultrasound evaluations of the scar will commence after the dermal scratch is completed and thereafter when the wound is healed (defined as >90% epithelialization of the wound with no exudate - approximately 1-3 weeks following wounding) and repeated on Day 20 (+/- 3), Day 27 (+/- 2), Day 48 (+/- 7) Day 76 (+/-14), Day 104 (+/- 15).

Two punch biopsies will be performed on the maximally thick region of each scar on Day 28 and day 104 for immunohistochemistry analysis of a-SMA (smooth muscle actin) and β-catenin, collagen orientation, and RT-qPCR analysis of type I and type III collagen, the β-catenin target gene (AXIN-2), TGF- β1 and decorin.

Subjects may request that the scar be completely excised on or after D104 under local anesthetic (1% xylocaine with epinephrine 1:100,000) and repaired using 4(0) monocril suture in the subcuticular plain to produce a fine linear scar. Tissue removed from this procedure will be used for immunohistochemistry analysis of β-catenin and RT-qPCR analysis of type I and type III collagen, the β-catenin target gene (AXIN-2), TGF- β1 and decorin.

Plan for Data Analysis:

All calculations and analyses will be performed using SAS version 9.4 or higher resident on the HP Unix (HPUX B.11.11 or higher. The continuous data will be summarized via PROC UNIVARIATE - mean, standard deviation, median, minimum, and maximum. The Safety Population will be used for analysis of adverse events, tolerability reactions, clinical evaluations, and laboratory tests. The ITT Population will be used for all other analyses.

For any assessments that are not performed per hip (e.g. adverse event reporting), results will be grouped by treatment (NEFOPAM 3.0% and placebo, placebo alone). For assessments that are performed separately on each hip (e.g. tolerability, POSAS scale), results will be grouped two ways: (1) By within-subject differences between hips grouped by the 3 treatment groups; and (2) By overall group mean value by treatment applied.

Tolerability is assessed separately for each hip by the investigator using a 5-point scale that ranges from 0 (No visible reaction) to 4 (Severe erythema with induration, vesicles or pustules and/or erosion/ulceration). While Likert scales are ordinal in nature, parametric methods are still robust and appropriate for analysis (43). Thus, for the assessment of tolerability, an ANCOVA model will be used to compare the within-subject difference between active and placebo hips (or, for placebo-only subjects, between left and right hips) in average tolerability. The average tolerability for each subject-hip will be calculated across all non-missing scheduled visits.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female burn, or trauma patients aged >18 - <65 years with 5-70% TBSA deep second or third degree burns who have uninjured skin in both the lateral hip regions and have voluntarily signed the Informed Consent Form (ICF).
2. Subjects with clinically acceptable results at screening for the laboratory tests specified in the trial protocol.
3. Women of childbearing potential must provide a negative pregnancy serum/urine test at time of screening and have to be compliant with an effective form of birth control throughout the entire study. Non-childbearing potential means subjects have had a history of tubal ligation or a hysterectomy or are post-menopausal with no menses for at least 1 year prior to enrolment in the study.
4. Subjects, who are, in the opinion of the Investigator, able to understand the study, co-operate with the study procedures and are willing to return to the clinic for all of the required follow-up visits.
5. Subjects must be able to cooperate with requirements of the study (e.g. able to speak, read and write English, and will be expected to be available for adverse event monitoring for the duration of the study).
6. Healthy subjects must have ALT and AST < 2 × ULN and TB < ULN at entry.
7. Subjects with carcinoma in situ or stage 1 cancer of the skin and other tissues will be acceptable once acceptable clinical management of the carcinoma has been established.
8. Patients who have well controlled HIV as defined by a viral load amount of HIV in the blood that is undetectable i.e. a: viral load less than 40 to 50 copies/ml and cannot be detected by standard tests for HIV, Hep B or Hep C will be included after consultation with an infectious disease expert.

Exclusion Criteria:

1. Currently Subjects involved any other intervention trial(s) where the intervention could possibly affect wound healing to be eligible for enrolment in the SCX-001 (Nefopam) Cream study.
2. Subjects who have scarring from previous interventions or evidence of thermal, electrical or radiation burn scars, tattoos, birthmarks or moles within 5 cm of the treatment site.
3. Exclusion criteria specific to burn patients in addition to the previously described factors would include severe inhalation injury requiring FiO2 >50%, renal failure requiring dialysis or hemodynamic instability requiring vasopressor therapy at the time of initiation of therapy.
4. Subjects with a history or family history of abnormal keloid scarring.
5. Subjects with additional concurrent illnesses or conditions that may have interfered with wound healing like neoplastic, immune-mediated, or primary infectious disease (e.g. carcinoma, vasculitis, connective tissue disease, immune system disorders, rheumatoid arthritis, chronic renal impairment, significant hepatic impairment, inadequately or uncontrolled congestive heart failure or diabetes mellitus) or any clinically significant medical condition or history of any condition which may impair wound healing.
6. Subjects with a skin disorder that is chronic or currently active and which the investigator considers will adversely affect the healing of acute wounds or will involve the areas to be examined in this trial (including psoriasis, dermatitis, eczema)
7. Subjects with a body mass index <15 or >35 kg/m2.
8. A history of radiotherapy to the study scar area.
9. Subjects who are positive for HIV, hepatitis B or C.
10. Subjects who have known sensitivities to SCX-001 (Nefopam) Cream, structurally related compounds or any of the constituents of SCX-001 (Nefopam) Cream.
11. Subjects who have known sensitivities to EMLA cream, chlorhexidine or adhesive dressings.
12. Elder patients (> 65 years), patients with epilepsy, patients with urinary retention, or or when administered with other anticholinergic or sympathomimetic drugs or monoamine oxidase inhibitors (MAOIs) or tricyclic antidepressants.
13. Subjects with end stage renal disease, where eGFR </= 30 mL/min.

    -

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of efficacy by measuring scar/wound area at day 1. | Digital photography of the wound/scar will be performed at day 1.
  To check the efficacy of the Nefopam cream all comparisons will be made between the Nefopam cream and the Placebo at different time point. Wound area will be measured using images obtained through digital photography on day 1 post operatively. Each image will be analyzed twice and the values averaged to provide an estimate of wound area (mm2) for each wound. Within-subject differences in wound area will be calculated and summarized by treatment group.
Assessment of efficacy by measuring scar/wound area at day 21. | Digital photography of the wound/scar will be performed at day 21.
  To check the efficacy of the Nefopam cream all comparisons will be made between the Nefopam cream and the Placebo at different time point. Wound area will be measured using images obtained through digital photography on day 1 post operatively. Each image will be analyzed twice and the values averaged to provide an estimate of wound area (mm2) for each wound. Within-subject differences in wound area will be calculated and summarized by treatment group.
Assessment of efficacy by measuring scar/wound area at day 27. | Digital photography of the wound/scar will be performed at day 27.
  To check the efficacy of the Nefopam cream all comparisons will be made between the Nefopam cream and the Placebo at different time point. Wound area will be measured using images obtained through digital photography on day 1 post operatively. Each image will be analyzed twice and the values averaged to provide an estimate of wound area (mm2) for each wound. Within-subject differences in wound area will be calculated and summarized by treatment group.
Assessment of efficacy by measuring scar/wound area at day 48. | Digital photography of the wound/scar will be performed at day 48.
  To check the efficacy of the Nefopam cream all comparisons will be made between the Nefopam cream and the Placebo at different time point. Wound area will be measured using images obtained through digital photography on day 1 post operatively. Each image will be analyzed twice and the values averaged to provide an estimate of wound area (mm2) for each wound. Within-subject differences in wound area will be calculated and summarized by treatment group.
Assessment of efficacy by measuring scar/wound area at day 76. | Digital photography of the wound/scar will be performed at day 76.
  To check the efficacy of the Nefopam cream all comparisons will be made between the Nefopam cream and the Placebo at different time point. Wound area will be measured using images obtained through digital photography on day 1 post operatively. Each image will be analyzed twice and the values averaged to provide an estimate of wound area (mm2) for each wound. Within-subject differences in wound area will be calculated and summarized by treatment group.
Assessment of efficacy by measuring scar/wound area at day 104. | Digital photography of the wound/scar will be performed at day 104.
  To check the efficacy of the Nefopam cream all comparisons will be made between the Nefopam cream and the Placebo at different time point. Wound area will be measured using images obtained through digital photography on day 1 post operatively. Each image will be analyzed twice and the values averaged to provide an estimate of wound area (mm2) for each wound. Within-subject differences in wound area will be calculated and summarized by treatment group.
Assessment of efficacy by measuring scar/wound depth at day 1. | Dermal ultrasound analysis of the wound/scar will be performed at day 1.
  To check the efficacy of the Nefopam cream all comparisons will be made between the Nefopam cream and the Placebo at different time point. At each visit there are three (3) measurements of wound depth at three (3) different points (deep end, mid-point, superficial end) will be taken. Scar depth will be measured in mm, based on ultrasound readings taken at scheduled assessment times.
Assessment of efficacy by measuring scar/wound depth at day 21. | Dermal ultrasound analysis of the wound/scar will be performed at day 21.
  To check the efficacy of the Nefopam cream all comparisons will be made between the Nefopam cream and the Placebo at different time point. At each visit there are three (3) measurements of wound depth at three (3) different points (deep end, mid-point, superficial end) will be taken. Scar depth will be measured in mm, based on ultrasound readings taken at scheduled assessment times.
Assessment of efficacy by measuring scar/wound depth at day 27. | Dermal ultrasound analysis of the wound/scar will be performed at day 27.
  To check the efficacy of the Nefopam cream all comparisons will be made between the Nefopam cream and the Placebo at different time point. At each visit there are three (3) measurements of wound depth at three (3) different points (deep end, mid-point, superficial end) will be taken. Scar depth will be measured in mm, based on ultrasound readings taken at scheduled assessment times.
Assessment of efficacy by measuring scar/wound depth at day 48. | Dermal ultrasound analysis of the wound/scar will be performed at day 48.
  To check the efficacy of the Nefopam cream all comparisons will be made between the Nefopam cream and the Placebo at different time point. At each visit there are three (3) measurements of wound depth at three (3) different points (deep end, mid-point, superficial end) will be taken. Scar depth will be measured in mm, based on ultrasound readings taken at scheduled assessment times.
Assessment of efficacy by measuring scar/wound depth at day 76. | Dermal ultrasound analysis of the wound/scar will be performed at day 76.
  To check the efficacy of the Nefopam cream all comparisons will be made between the Nefopam cream and the Placebo at different time point. At each visit there are three (3) measurements of wound depth at three (3) different points (deep end, mid-point, superficial end) will be taken. Scar depth will be measured in mm, based on ultrasound readings taken at scheduled assessment times.
Assessment of efficacy by measuring scar/wound depth at day 104. | Dermal ultrasound analysis of the wound/scar will be performed at day 104.
  To check the efficacy of the Nefopam cream all comparisons will be made between the Nefopam cream and the Placebo at different time point. At each visit there are three (3) measurements of wound depth at three (3) different points (deep end, mid-point, superficial end) will be taken. Scar depth will be measured in mm, based on ultrasound readings taken at scheduled assessment times.
Assessment of efficacy by measuring scar erythema and pigmentation at day 1. | Mexameter® assessments of the wound/scar will be performed at day 1.
  To check the efficacy of the Nefopam cream all comparisons will be made between the Nefopam cream and the Placebo at different time point.
  Once the wound has been determined to be closed, Mexameter® assessments will be performed at scheduled visits to check scar erythema and pigmentation . Mexameter® assessments will be performed at three standardized positions along each scar. At each position, three individual measurements will be taken and the mean and standard deviation will be determined for both erythema and pigmentation at each of the three measurement positions.
Assessment of efficacy by measuring scar erythema and pigmentation at day 21. | Mexameter® assessments of the wound/scar will be performed at day 21.
  To check the efficacy of the Nefopam cream all comparisons will be made between the Nefopam cream and the Placebo at different time point.
  Once the wound has been determined to be closed, Mexameter® assessments will be performed at scheduled visits to check scar erythema and pigmentation . Mexameter® assessments will be performed at three standardized positions along each scar. At each position, three individual measurements will be taken and the mean and standard deviation will be determined for both erythema and pigmentation at each of the three measurement positions.
Assessment of efficacy by measuring scar erythema and pigmentation at day 27. | Mexameter® assessments of the wound/scar will be performed at day 27.
  To check the efficacy of the Nefopam cream all comparisons will be made between the Nefopam cream and the Placebo at different time point.
  Once the wound has been determined to be closed, Mexameter® assessments will be performed at scheduled visits to check scar erythema and pigmentation . Mexameter® assessments will be performed at three standardized positions along each scar. At each position, three individual measurements will be taken and the mean and standard deviation will be determined for both erythema and pigmentation at each of the three measurement positions.
Assessment of efficacy by measuring scar erythema and pigmentation at day 48. | Mexameter® assessments of the wound/scar will be performed at day 48.
  To check the efficacy of the Nefopam cream all comparisons will be made between the Nefopam cream and the Placebo at different time point.
  Once the wound has been determined to be closed, Mexameter® assessments will be performed at scheduled visits to check scar erythema and pigmentation . Mexameter® assessments will be performed at three standardized positions along each scar. At each position, three individual measurements will be taken and the mean and standard deviation will be determined for both erythema and pigmentation at each of the three measurement positions.
Assessment of efficacy by measuring scar erythema and pigmentation at day 76. | Mexameter® assessments of the wound/scar will be performed at day 76.
  To check the efficacy of the Nefopam cream all comparisons will be made between the Nefopam cream and the Placebo at different time point.
  Once the wound has been determined to be closed, Mexameter® assessments will be performed at scheduled visits to check scar erythema and pigmentation . Mexameter® assessments will be performed at three standardized positions along each scar. At each position, three individual measurements will be taken and the mean and standard deviation will be determined for both erythema and pigmentation at each of the three measurement positions.
Assessment of efficacy by measuring scar erythema and pigmentation at day 104. | Mexameter® assessments of the wound/scar will be performed at day 104.
  To check the efficacy of the Nefopam cream all comparisons will be made between the Nefopam cream and the Placebo at different time point.
  Once the wound has been determined to be closed, Mexameter® assessments will be performed at scheduled visits to check scar erythema and pigmentation . Mexameter® assessments will be performed at three standardized positions along each scar. At each position, three individual measurements will be taken and the mean and standard deviation will be determined for both erythema and pigmentation at each of the three measurement positions.
Assessment of efficacy by assessing scar/wound healing at day 6 (during Nefopam cream treatment). | Wound healing will be measured at day 6 (during Nefopam cream treatment).
  Wound healing, defined as 100% epithelialization of the wound with no exudate. Percentage of wounds healed by visit by treatment will be summarized. The difference in proportions of healed wounds will be calculated within treatment group (active treatment against placebo within that group).
Assessment of efficacy by assessing scar/wound healing at day 13 (during Nefopam cream treatment). | Wound healing will be measured at day 13 (during Nefopam cream treatment).
  Wound healing, defined as 100% epithelialization of the wound with no exudate. Percentage of wounds healed by visit by treatment will be summarized. The difference in proportions of healed wounds will be calculated within treatment group (active treatment against placebo within that group).
Assessment of efficacy by assessing scar/wound healing at day 20 (during Nefopam cream treatment). | Wound healing will be measured at day 20 (during Nefopam cream treatment).
  Wound healing, defined as 100% epithelialization of the wound with no exudate. Percentage of wounds healed by visit by treatment will be summarized. The difference in proportions of healed wounds will be calculated within treatment group (active treatment against placebo within that group).
Assessment of efficacy by assessing scar/wound healing at day 27 (after completion of Nefopam cream application). | Wound healing will be measured at day 27 (after completion of Nefopam cream application).
  Wound healing, defined as 100% epithelialization of the wound with no exudate. Percentage of wounds healed by visit by treatment will be summarized. The difference in proportions of healed wounds will be calculated within treatment group (active treatment against placebo within that group).
Assessment of efficacy by assessing scar/wound healing at day 48 (after completion of Nefopam cream application). | Wound healing will be measured at day 48 (after completion of Nefopam cream application).
  Wound healing, defined as 100% epithelialization of the wound with no exudate. Percentage of wounds healed by visit by treatment will be summarized. The difference in proportions of healed wounds will be calculated within treatment group (active treatment against placebo within that group).
Assessment of efficacy by assessing scar/wound healing at day 104 (after completion of Nefopam cream application). | Wound healing will be measured at day 104 (after completion of Nefopam cream application).
  Wound healing, defined as 100% epithelialization of the wound with no exudate. Percentage of wounds healed by visit by treatment will be summarized. The difference in proportions of healed wounds will be calculated within treatment group (active treatment against placebo within that group).
Assessment of the scar using the Patient and Observer Scar Assessment Scales (POSAS) at day 27 (after completion of Nefopam cream application). | Patient and Observer Scar Assessment Scales (POSAS) will be performed at day 27 (after completion of Nefopam cream application).
  The POSAS consists of a section completed by the subject and sections completed by three observers - once for each hip, at each post-wound-closure visit. The Patient section consists of seven (7) questions on 10-point scales regarding scar pain, itchiness, colour, stiffness, thickness, irregularity, and an overall assessment. The Observer sections consist of seven (7) 10-point scales regarding vascularity, pigmentation, thickness, relief, pliability, surface area, and overall assessment.
  On Y axis POSAS scoring will be taken and on X axis outcome from the patients at different time point will be recorded. Each of the seven questions has a 10-point scoring system, with 1 representing normal skin and 10 the worst imaginable scar or sensation. The total score of both scales consists of adding the scores of each of the seven questions (range, 7 to 70). The lowest score, 7, reflects normal skin, whereas the highest score, 70, reflects the worst imaginable scar.
Assessment of the scar using the Patient and Observer Scar Assessment Scales (POSAS) at day 48 (after completion of Nefopam cream application). | Patient and Observer Scar Assessment Scales (POSAS) will be performed at day 48 (after completion of Nefopam cream application).
  The POSAS consists of a section completed by the subject and sections completed by three observers - once for each hip, at each post-wound-closure visit. The Patient section consists of seven (7) questions on 10-point scales regarding scar pain, itchiness, colour, stiffness, thickness, irregularity, and an overall assessment. The Observer sections consist of seven (7) 10-point scales regarding vascularity, pigmentation, thickness, relief, pliability, surface area, and overall assessment.
  On Y axis POSAS scoring will be taken and on X axis outcome from the patients at different time point will be recorded. Each of the seven questions has a 10-point scoring system, with 1 representing normal skin and 10 the worst imaginable scar or sensation. The total score of both scales consists of adding the scores of each of the seven questions (range, 7 to 70). The lowest score, 7, reflects normal skin, whereas the highest score, 70, reflects the worst imaginable scar.
Assessment of the scar using the Patient and Observer Scar Assessment Scales (POSAS) at day 76 (after completion of Nefopam cream application). | Patient and Observer Scar Assessment Scales (POSAS) will be performed at day 76 (after completion of Nefopam cream application).
  The POSAS consists of a section completed by the subject and sections completed by three observers - once for each hip, at each post-wound-closure visit. The Patient section consists of seven (7) questions on 10-point scales regarding scar pain, itchiness, colour, stiffness, thickness, irregularity, and an overall assessment. The Observer sections consist of seven (7) 10-point scales regarding vascularity, pigmentation, thickness, relief, pliability, surface area, and overall assessment.
  On Y axis POSAS scoring will be taken and on X axis outcome from the patients at different time point will be recorded. Each of the seven questions has a 10-point scoring system, with 1 representing normal skin and 10 the worst imaginable scar or sensation. The total score of both scales consists of adding the scores of each of the seven questions (range, 7 to 70). The lowest score, 7, reflects normal skin, whereas the highest score, 70, reflects the worst imaginable scar.
Assessment of the scar using the Patient and Observer Scar Assessment Scales (POSAS) at day 104 (after completion of Nefopam cream application). | Patient and Observer Scar Assessment Scales (POSAS) will be performed at day 104 (after completion of Nefopam cream application).
  The POSAS consists of a section completed by the subject and sections completed by three observers - once for each hip, at each post-wound-closure visit. The Patient section consists of seven (7) questions on 10-point scales regarding scar pain, itchiness, colour, stiffness, thickness, irregularity, and an overall assessment. The Observer sections consist of seven (7) 10-point scales regarding vascularity, pigmentation, thickness, relief, pliability, surface area, and overall assessment.
  On Y axis POSAS scoring will be taken and on X axis outcome from the patients at different time point will be recorded. Each of the seven questions has a 10-point scoring system, with 1 representing normal skin and 10 the worst imaginable scar or sensation. The total score of both scales consists of adding the scores of each of the seven questions (range, 7 to 70). The lowest score, 7, reflects normal skin, whereas the highest score, 70, reflects the worst imaginable scar.
Assessment of efficacy by performing qPCR of the fibrotic molecules at day 27 (after completion of Nefopam cream application). | Two punch biopsies will be performed on the maximally thick region of each scar on Day 27 (after completion of Nefopam cream application).
  To determine the efficacy of Nefopam cream versus placebo on the fibrotic molecules including type I and type III collagen, β-catenin target gene (AXIN-2), TGF- β1, and decorin, quantitative measures will be performed. TGF-β1, AXIN-2, decorin, and collagen types I and III will be expressed as fold-change values; fold change values will be calculated based on the double delta Ct method (where fold change = 2-∆∆CT).
Assessment of efficacy by performing qPCR of the fibrotic molecules at day 104(after completion of Nefopam cream application). | Two punch biopsies will be performed on the maximally thick region of each scar on Day 104 (after completion of Nefopam cream application).
  To determine the efficacy of Nefopam cream versus placebo on the fibrotic molecules including type I and type III collagen, β-catenin target gene (AXIN-2), TGF- β1, and decorin, quantitative measures will be performed. TGF-β1, AXIN-2, decorin, and collagen types I and III will be expressed as fold-change values; fold change values will be calculated based on the double delta Ct method (where fold change = 2-∆∆CT).
Assessment of efficacy by performing Immunohistochemistry at day 27(after completion of Nefopam cream application). | Two punch biopsies will be performed on the maximally thick region of each scar on Day 27 (after completion of Nefopam cream application).
  To determine the efficacy of Nefopam cream versus placebo, protein expression of fibrotic molecules will be measured by immunohistochemistry.
  a-SMA (smooth muscle actin) and β -catenin immunohistochemistry will be performed at day 27.
Assessment of efficacy by performing Immunohistochemistry at day 104 (after completion of Nefopam cream application). | Two punch biopsies will be performed on the maximally thick region of each scar on Day 104 (after completion of Nefopam cream application).
  To determine the efficacy of Nefopam cream versus placebo, protein expression of fibrotic molecules will be measured by immunohistochemistry. a-SMA (smooth muscle actin) and β -catenin immunohistochemistry will be performed at day 104.

SECONDARY OUTCOMES:
Assessment of Safety by assessing drug tolerability. | Treatment tolerability will be assessed regularly during the first 21 days of the trial.
  At each clinic visit the area surrounding each wound/scar where the study drug had been applied will be assessed for tolerability using the following validated scoring assessment:
  0 = no visible reaction,
  1. = faint, minimal erythema,
  2. = erythema,
  3. = erythema with induration or vesicles,
  4. = severe erythema with induration, vesicles or bullae or pustules and/or erosion/ulceration.
  Using an ANCOVA model, estimated average difference in average tolerability across scheduled visits will be calculated between active and placebo hips with treatment differences and 95% confidence intervals. These results of mean within-subject difference between hips will be presented by treatment group.
Assessment of heart rate. | Hear rate will be measured at day 27, 76, and 104.
  Heart rate will be assessed and summarized as mean values with variance, including the change from baseline, by treatment group at each scheduled time point.
  (PS: However data will be presented as mean value and variance, but unit will be the same, as we are measuring only one outcome here (heart rate) ).
Assessment of temperature. | Body temperature will be measured at day 27, 76, and 104.
  Body temperature will be assessed and summarized as mean values with variance, including the change from baseline, by treatment group at each scheduled time point.
  (PS: However data will be presented as mean value and variance, but unit will be the same, as we are measuring only one outcome here (body temperature) ).
Assessment of blood pressure. | Blood pressure will be measured at day 27, 76, and 104.
  Blood pressure (systolic and diastolic) will be assessed and summarized as mean values with variance, including the change from baseline, by treatment group at each scheduled time point.
  (PS: However data will be presented as mean value and variance, but unit will be the same, as we are measuring only one outcome here (blood pressure) ).
Assessment of respiration. | Respiration will be measured at day 27, 76, and 104.
  Respiration will be assessed and summarized as mean values with variance, including the change from baseline, by treatment group at each scheduled time point.
  (PS: However data will be presented as mean value and variance, but unit will be the same, as we are measuring only one outcome here).
Measurement of routine hematology parameters. | Routine hematology parameters will be measured at day 27, 76 and 104.
  Routine hematology parameters like CBC (complete blood count); (CBC is a group of tests that evaluate the cells that circulate in blood, including red blood cells (RBCs), white blood cells (WBCs), and platelets (PLTs), HB (hemoglobin) , HCT (hematocrit), FIB (fibrinogen) will be presented as mean values with variability and change (absolute and relative) from baseline for each laboratory parameter at each scheduled time point.
  (There are multiple assessments but they all come in one outcome measure (hematology parameters). We can put them separately but as they all come together, when we refer to hematology test. It will make more sense to the study, if we put them together. Second these test are the routine checkup for the participants ).
Measurement of routine clinical chemistry parameters. | Routine clinical chemistry parameters will be measured at day 27, 76 and 104.
  Routine Clinical chemistry parameters like GLUCF (glucose-fasting), GLUCP (glucose, 2 hour, post cibum), Na (sodium), K (potassium), CL (chloride), CREA (creatinine), CA (calcium), ALB (albumin), ALP (alk phos), LDL (low-density lipoproteins), HDL (high-density lipoprotein), TRIG (triglycerides), CHOL (cholesterol) will be presented as mean values with variability and change (absolute and relative) from baseline for each laboratory parameter at each scheduled time point.
  (There are multiple assessments but they all come in one outcome measure (hematology parameters). We can put them separately but as they all come together, when we refer to hematology test. It will make more sense to the study, if we put them together. Second these test are the routine checkup for the participants ).
Serum Nefopam absorption assessment. | Serum Nefopam analysis will be carried out at time zero, 8 hours and 24 hours after initiation of the treament.
  Serum Nefopam levels will be measured in the first five patients at time 0 (before application of the drug), 8 hours (after initiation of the first day treatment) and 24 hours (after initiation of the first day treatment) to check concentration of Nefopam.

CONTACTS AND LOCATIONS:
Overall Officials: Edward E Tredget, MD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Case MT, Smith JK, Nelson RA. Reproductive, acute and subacute toxicity studies with nefopam in laboratory animals. Toxicol Appl Pharmacol. 1975 Jul;33(1):46-51. doi: 10.1016/0041-008x(75)90242-2. No abstract available. PMID 1162704
- [Background] Dunkin CSJ, Pleat JM, Gillespie PH, Tyler MPH, Roberts AHN, McGrouther DA. Scarring occurs at a critical depth of skin injury: precise measurement in a graduated dermal scratch in human volunteers. Plast Reconstr Surg. 2007 May;119(6):1722-1732. doi: 10.1097/01.prs.0000258829.07399.f0. PMID 17440346
- [Background] Honardoust D, Varkey M, Marcoux Y, Shankowsky HA, Tredget EE. Reduced decorin, fibromodulin, and transforming growth factor-beta3 in deep dermis leads to hypertrophic scarring. J Burn Care Res. 2012 Mar-Apr;33(2):218-27. doi: 10.1097/BCR.0b013e3182335980. PMID 22079916
- [Background] Poon R, Hong H, Wei X, Pan J, Alman BA. A high throughput screen identifies Nefopam as targeting cell proliferation in beta-catenin driven neoplastic and reactive fibroproliferative disorders. PLoS One. 2012;7(5):e37940. doi: 10.1371/journal.pone.0037940. Epub 2012 May 30. PMID 22666417
- [Background] Case MT, Smith JK, Nelson RA. Chronic oral toxicity studies of nefopam hydrochloride in rats and dogs. Toxicol Appl Pharmacol. 1976 May;36(2):301-6. doi: 10.1016/0041-008x(76)90009-0. No abstract available. PMID 1273848
- [Background] Mather GG, Labroo R, Le Guern ME, Lepage F, Gillardin JM, Levy RH. Nefopam enantiomers: preclinical pharmacology/toxicology and pharmacokinetic characteristics in healthy subjects after intravenous administration. Chirality. 2000 Mar;12(3):153-9. doi: 10.1002/(SICI)1520-636X(2000)12:33.0.CO;2-V. PMID 10689295